CLINICAL TRIAL: NCT02457247
Title: A Randomized, Open-Label, 2-Way Cross-Over, Phase 4 Study to Evaluate Subject Preference and Acceptability of a New Formulation of Calcichew D3 in Adult Patients Eligible for Calcium and Vitamin D Supplementation
Brief Title: Calcichew D3 Preference Study in Participants Eligible for Calcium and Vitamin D Supplementation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Calcichew-4001; 2014-005619-18 (EudraCT Number); U1111-1166-8818 (Registry Identifier: WHO); 15/NW/0275 (Registry Identifier: NRES)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-08

CONDITIONS: Calcium and Vitamin D Deficiencies
Keywords: Drug therapy
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test Group 1: Sequence AB (Experimental): Calcichew D3 500/400 (Calcium 500 mg/400 IU Vitamin D3) [A], chewable tablets, orally, twice, daily, on Days 1 through 14, followed by Adcal-D3 (Calcium 600 mg / 400 IU Vitamin D3) [B], chewable tablets, orally, twice, daily, on Days 15 through 28.
  Interventions: Drug: Calcichew D3; Drug: Adcal-D3
- Test Group 1: Sequence BA (Experimental): Adcal-D3 (Calcium 600 mg / 400 IU Vitamin D3), chewable tablets, orally, twice, daily, on Days 1 through 14, followed by, Calcichew D3 500/400 (Calcium 500 mg/400 IU Vitamin D3), chewable tablets, orally, twice, daily, on Days 15 through 28.
  Interventions: Drug: Calcichew D3; Drug: Adcal-D3
- Test Group 2: Sequence CD (Experimental): Calcichew D3 500/800 (Calcium 500 mg/800 IU Vitamin D3) [C], chewable tablets, orally, once, daily, on Days 1 through 14, followed by Kalcipos-D (Calcium 500 mg/800 IU Vitamin D3) [D], chewable tablets, orally, once, daily, on Days 15 through 28.
  Interventions: Drug: Calcichew D3; Drug: Kalcipos-D
- Test Group 2: Sequence DC (Experimental): Kalcipos-D (Calcium 500 mg/800 IU Vitamin D3), chewable tablets, orally, once, daily, on Days 1 through 14, followed by, Calcichew D3 500/800 (Calcium 500 mg/800 IU Vitamin D3), chewable tablets, orally, once, daily, on Days 15 through 28.
  Interventions: Drug: Calcichew D3; Drug: Kalcipos-D

INTERVENTIONS:
Drug: Calcichew D3 — Calcichew D3 500/400 (Calcium 500 mg/400 IU Vitamin D3) Calcichew D3 500/800 (Calcium 500 mg/800 IU Vitamin D3)
Drug: Adcal-D3 — Adcal-D3 (Calcium 600mg/400 IU Vitamin D3)
  Arms: Test Group 1: Sequence AB; Test Group 1: Sequence BA
Drug: Kalcipos-D — Kalcipos-D (Calcium 500mg/800 IU Vitamin D3)
  Arms: Test Group 2: Sequence CD; Test Group 2: Sequence DC

SUMMARY:
The purpose of this study is to compare the preference of Calcichew D3 500/400 (containing 500 mg calcium and 400 IU of vitamin D) with Adcal-D3 600/400 (containing 600 mg of calcium and 400 IU of vitamin D) in Test Group 1, and to compare Calcichew D3 500/800 (containing 500 mg calcium and 800 IU vitamin D) with Kalcipos-D 500/800 (containing 500 mg of calcium and 800 IU of vitamin D) in Test Group 2.

DETAILED DESCRIPTION:
The drug being tested in this study is called Calcichew D3 new formulations: Calcichew D3 500/400 and Calcichew D3 500/800. Calcichew D3 500/400 and Calcichew D3 500/800 are being tested to treat or prevent calcium or vitamin D deficiencies. Calcichew D3 500/400 will be compared to Adcal-D3 600/400 as prescribed in clinical practice and Calcichew D3 500/800 will be compared to Kalcipos-D 500/800 as prescribed in clinical practice.

This Crossover study will enroll approximately 276 patients equally divided between the two test groups (138 patients each). Within each test group, participants will be randomly assigned (by chance, like flipping a coin) to one of two treatment sequences, as described below.

Test Group 1:

* Calcichew D3 500/400 (containing 500 mg calcium and 400 IU of vitamin D) chewable tablet
* Adcal-D3 600/400 (containing 600 mg of calcium and 400 IU of vitamin D) chewable tablet

Test Group 2:

* Calcichew D3 500/800 (containing 500 mg calcium and 800 IU vitamin D) chewable tablets
* Kalcipos-D 500/800 (containing 500 mg of calcium and 800 IU of vitamin D) chewable tablets

Participants in Test Group 1 will take either Calcichew D3 500/400 or Adcal-D3 600/400 for 14 days and then will crossover to take either Calcichew D3 500/400 or Adcal-D3 600/400 treatment for 14 days. Participants in Test Group 2 will take either Calcichew D3 500/800 or Kalcipos-D 600/400 for 14 days and then will crossover to take either Calcichew D3 500/800 or Kalcipos-D treatment for 14 days.

This multi-center trial will be conducted In the United Kingdom and Germany. The overall time to participate in this study is 28 days. Participants will make multiple visits to the clinic including a final visit assessment at Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Is eligible for or currently receiving treatment with calcium and vitamin D supplement as determined by the treating clinician in accordance with local treatment guidelines.
4. Eligible participants will either be:

   1. Aged 65 years or older requiring calcium and vitamin D supplementation for the prevention or treatment of deficiencies, or
   2. Aged 18 years or older that require calcium and vitamin D as an adjunct to specific osteoporosis treatment in participants at risk of calcium and vitamin D deficiencies.
5. Is male or female.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study, and for 12 weeks after last dose of study medication.

Exclusion Criteria:

1. Has received Calcichew D3, Adcal-D3 (if the participant is in Test Group 1) or Kalcipos-D (if the participant is in Test Group 2) within the 6 months prior to the first dose of study medication.
2. Has received any investigational compound within 30 days prior to Screening.
3. Has a disease and/or condition resulting in hypercalcaemia and/or hypercalciuria and for which the study drugs are contraindicated e.g. Zollinger-Ellison syndrome, nephrolithiasis.
4. Has any of the contraindications listed in the corresponding Summary of Product Characteristics (SPC) of the study drug that the participant may receive depending on the Test Group: Calcichew D3 or Adcal-D3 (if the participant is in Test Group 1); Calcichew D3 or Kalcipos-D (if the participant is in Test Group 2).
5. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
6. Has a history of hypersensitivity or allergies to the active substances or to any of the excipients in the investigational products.
7. Has a history of known fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency.
8. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 12 weeks after participating in this study; or intending to donate ova during such time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (9):
- Germany (4):
  - Berlin
  - Bochum
  - Frankfurt
  - Leipzig
- United Kingdom (5):
  - Reading, Berkshire
  - Birmingham
  - Chorley
  - Liverpool
  - Manchester

REFERENCES:
- [Derived] Thomasius F, Keung Nip T, Ivan P. Phase IV randomized preference study in patients eligible for calcium and vitamin D supplementation. Curr Med Res Opin. 2016 Oct;32(10):1623-1631. doi: 10.1080/03007995.2016.1202817. Epub 2016 Jun 29. PMID 27322906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in the United Kingdom and Germany from 02 June 2015 to 27 August 2015.
Pre-assignment Details: Participants eligible for Vitamin D and Calcium supplements were enrolled equally in 1 of 2 Test Groups to determine the preference between 2 treatments.
  Group 1: Calcichew D3 500/400 and Adcal-D3 600/400 or Group 2: Calcichew D3 500/800 and Kalcipos-D 500/800.
Period: Period 1
Arm/Group | Test Group 1: Sequence AB | Test Group 1: Sequence BA | Test Group 2: Sequence CD | Test Group 2: Sequence DC
Started | 68 | 70 | 68 | 70
Completed | 66 | 68 | 68 | 70
Not Completed | 2 | 2 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 0 | 1 | 0 | 0
Not completed — Significant Protocol Deviation | 1 | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Test Group 1: Sequence AB | Test Group 1: Sequence BA | Test Group 2: Sequence CD | Test Group 2: Sequence DC
Started | 66 | 68 | 68 | 70
Completed | 64 | 65 | 68 | 70
Not Completed | 2 | 3 | 0 | 0
Not completed — Pretreatment Event/Adverse Event | 0 | 1 | 0 | 0
Not completed — Significant Protocol Deviation | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Voluntary Withdrawal | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group 1: Sequence AB | Test Group 1: Sequence BA | Test Group 2: Sequence CD | Test Group 2: Sequence DC | Total
Number analyzed (Participants) | 68 | 70 | 68 | 70 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (7.37) [65 to 80] | 70.8 (4.94) [65 to 85] | 70.9 (7.37) [36 to 85] | 69.9 (7.03) [46 to 84] | NA (NA) [36 to 85] — Test Group 1 and Test Group 2 were analyzed separately for their respective region (UK and Germany, respectively); therefore, Total Mean and Standard Deviation are not available.
Age, Customized [Number; unit: participants]
  <65 years | 0 | 0 | 8 | 11 | 19
  ≥65 years | 68 | 70 | 60 | 59 | 257
Age, Customized [Number; unit: participants]
  Adults (18-64 Years) | 0 | 0 | 8 | 11 | 19
  From 65-84 Years | 68 | 69 | 58 | 59 | 254
  85 Years and Over | 0 | 1 | 2 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 60 | 60 | 201
  Male | 28 | 29 | 8 | 10 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 3 | 0 | 1 | 5
  Multiracial | 0 | 1 | 0 | 0 | 1
  White | 67 | 66 | 68 | 69 | 270
Region of Enrollment [Number; unit: participants]
  United Kingdom | 68 | 70 | 0 | 0 | 138
  Germany | 0 | 0 | 68 | 70 | 138
Height [Mean (Standard Deviation); unit: cm] — Height data is available for 65, 70, 68 and 70 participants, respectively.
  cm | 164.4 (7.44) [150 to 183] | 165.4 (8.95) [150 to 188] | 164.0 (7.73) [148 to 186] | 164.8 (7.78) [150 to 186] | NA (NA) [148 to 188] — Test Group 1 and Test Group 2 were analyzed separately for their respective region (UK and Germany, respectively); therefore, Total Mean and Standard Deviation are not available.
Weight [Mean (Standard Deviation); unit: kg] | 78.92 (15.383) [46.2 to 110.0] | 81.72 (23.559) [54.5 to 172.5] | 71.44 (13.799) [53.0 to 114.4] | 73.61 (16.340) [41.9 to 125.0] | NA (NA) [41.9 to 172.5] — Test Group 1 and Test Group 2 were analyzed separately for their respective region (UK and Germany, respectively); therefore, Total Mean and Standard Deviation are not available.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data is available for 65, 70, 68 and 70 participants, respectively.
  kg/m^2 | 29.157 (4.7766) [17.39 to 39.92] | 29.588 (6.5710) [19.92 to 55.52] | 26.478 (4.2362) [19.94 to 39.45] | 27.002 (5.1081) [17.96 to 46.48] | NA (NA) [17.39 to 55.52] — Test Group 1 and Test Group 2 were analyzed separately for their respective region (UK and Germany, respectively); therefore, Total Mean and Standard Deviation are not available.
BMI Categorical [Number; unit: participants]
  <25 kg/m^2 | 11 | 17 | 30 | 27 | 85
  25 to <30 kg/m^2 | 30 | 29 | 27 | 27 | 113
  ≥30 kg/m^2 | 24 | 24 | 11 | 16 | 75
  Missing | 3 | 0 | 0 | 0 | 3
Smoking Status [Number; unit: participants]
  Never Smoked | 28 | 31 | 41 | 35 | 135
  Ex-smoker | 32 | 33 | 18 | 24 | 107
  Current Smoker | 8 | 6 | 9 | 11 | 34
Alcohol Status [Number; unit: participants]
  Never Drank | 11 | 14 | 10 | 12 | 47
  Ex-drinker | 4 | 10 | 5 | 2 | 21
  Current Drinker | 53 | 46 | 53 | 56 | 208
History of Osteoporosis [Number; unit: participants]
  Yes | 1 | 3 | 28 | 24 | 56
  No | 67 | 67 | 40 | 46 | 220
History of Osteopenia [Number; unit: participants]
  Yes | 7 | 3 | 7 | 12 | 29
  No | 61 | 67 | 61 | 58 | 247
History of Fractures in the Last 10 Years [Number; unit: participants]
  Yes | 11 | 10 | 7 | 8 | 36
  No | 57 | 60 | 61 | 62 | 240

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Preference for Each Treatment Within Each Test Group
Description: Preference was assessed by a 3 box questionnaire. Participants checked off one of the boxes: I prefer the first product that was tested, I prefer the second product that was tested or I have no preference. Test Group 1 (United Kingdom): Calcichew D3 is 500/400 and the comparator is Adcal-D3. Test Group 2 (Germany): Calcichew D3 is 500/800 and the comparator is Kalcipos-D.
Time Frame: Day 28
Population: All randomized participants from the Full Analysis Set (FAS) who received at least 1 dose of study medication and responded to the preference questionnaire.
Measure: Number; unit: percentage of participants
Groups:
- Test Group 1: Total: Calcichew D3 500/400 (Calcium 500 mg/400 IU Vitamin D3) [A], chewable tablets, orally, twice, daily, for 14 days in either Period 1 or 2 and Adcal-D3 (Calcium 600 mg / 400 IU Vitamin D3) [B], chewable tablets, orally, twice, daily, for 14 days in either Period 1 or 2.
- Test Group 2: Total: Calcichew D3 500/800 (Calcium 500 mg/800 IU Vitamin D3) [C], chewable tablets, orally, once, daily, for 14 days in either Period 1 or 2 and Kalcipos-D (Calcium 500 mg/800 IU Vitamin D3) [D], chewable tablets, orally, for 14 days in either Period 1 or 2.
Arm/Group | Test Group 1: Sequence AB | Test Group 1: Sequence BA | Test Group 2: Sequence CD | Test Group 2: Sequence DC | Test Group 1: Total | Test Group 2: Total
Number analyzed (Participants) | 64 | 65 | 68 | 70 | 129 | 138
percentage of participants
  Preference for Calcichew D3 | 67.2 | 72.3 | 61.8 | 52.9 | 69.8 | 57.2
  Preference for Comparator | 28.1 | 12.3 | 29.4 | 37.1 | 20.2 | 33.3
  No Preference | 4.7 | 15.4 | 8.8 | 10.0 | 10.1 | 9.4

2. Secondary Outcome: Product Acceptability After Each 14 Day Dosing Period Within Each Test Group
Description: Product acceptability was assessed by a 6 item questionnaire evaluating the characteristics of the product: gritty, chalky, sweet, ease of chew, ease of swallow and sticky. Using a 100 mm visual analog scale (VAS) the participant put a vertical line through each horizontal line that best describes their level of agreement with each item using a 0 to 100 scale where: 0=far left of the line (best) to 100= far right of the line (worst). Linear mixed model was used for analysis with treatment and period as fixed effects and participants as a random effect.
Time Frame: Day 14 and Day 28
Population: The FAS included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mm
Groups:
- United Kingdom: Calcichew D3 500/400: Calcichew D3 500/400 (Calcium 500 mg/400 IU Vitamin D3) [A], chewable tablets, orally, twice, daily, on Days 1 through 14 or Days 15 through 28.
- United Kingdom: Adcal-D3: Adcal-D3 (Calcium 600 mg / 400 IU Vitamin D3), chewable tablets, orally, twice, daily, on Days 1 through 14 or Days 15 through 28.
- Germany: Calcichew D3 500/800: Calcichew D3 500/800 (Calcium 500 mg/800 IU Vitamin D3) [C], chewable tablets, orally, once, daily, on Days 1 through 14 or Days 15 through 28.
- Germany: Kalcipos-D: Kalcipos-D (Calcium 500 mg/800 IU Vitamin D3), chewable tablets, orally, once, daily, on Days 1 through 14 or Days 15 through 28.
Arm/Group | United Kingdom: Calcichew D3 500/400 | United Kingdom: Adcal-D3 | Germany: Calcichew D3 500/800 | Germany: Kalcipos-D
Number analyzed (Participants) | 138 | 138 | 138 | 138
mm
  Gritty | 19.2 (2.18) | 24.6 (2.18) | 28.4 (2.28) | 27.0 (2.28)
  Chalky | 23.2 (2.49) | 41.1 (2.49) | 25.9 (2.43) | 29.9 (2.43)
  Sweet/Bitter | 32.5 (1.74) | 34.5 (1.74) | 34.1 (1.67) | 38.0 (1.67)
  Chew | 8.1 (1.62) | 18.1 (1.62) | 12.2 (1.77) | 19.0 (1.78)
  Swallow | 10.8 (2.01) | 20.5 (2.00) | 11.0 (1.88) | 19.5 (1.89)
  Sticky | 6.1 (1.22) | 10.9 (1.22) | 8.2 (1.16) | 8.4 (1.16)

3. Secondary Outcome: Product Tolerability Expressed as the Percentage of Participants Who Experience at Least One Treatment-Emergent Adverse Event Within Each Test Group
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 to Day 28
Population: The Safety Analysis Set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | United Kingdom: Calcichew D3 500/400 | United Kingdom: Adcal-D3 | Germany: Calcichew D3 500/800 | Germany: Kalcipos-D
Number analyzed (Participants) | 135 | 136 | 138 | 138
percentage of participants | 14.8 | 9.6 | 5.1 | 4.3

ADVERSE EVENTS:
Time Frame: From first dose of the study drug to the last dose of study drug (Up to 28 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
  Safety Set included all participants who received at least 1 dose of study drug.
Arm/Group | United Kingdom: Calcichew D3 500/400 | United Kingdom: Adcal-D3 | Germany: Calcichew D3 500/800 | Germany: Kalcipos-D
Serious Adverse Events (participants affected / at risk) | 1/135 | 0/136 | 0/138 | 0/138
Other Adverse Events (participants affected / at risk) | 1/135 | 5/136 | 0/138 | 0/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | United Kingdom: Calcichew D3 500/400 (N=135) | United Kingdom: Adcal-D3 (N=136) | Germany: Calcichew D3 500/800 (N=138) | Germany: Kalcipos-D (N=138)
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | United Kingdom: Calcichew D3 500/400 (N=135) | United Kingdom: Adcal-D3 (N=136) | Germany: Calcichew D3 500/800 (N=138) | Germany: Kalcipos-D (N=138)
Constipation (Gastrointestinal disorders) | 1 | 5 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.